CLINICAL TRIAL: NCT07320053
Title: Effect of Longitudinal Care in Primary Health Care: An Analysis From the Patient's Perspective
Acronym: CUALIPRIM
Status: Completed | Type: Observational
Sponsor: IBS Granada (Other)
Collaborators: Universidad de Granada (Other); La Sociedad Española de Médicos de Atención Primaria (Other)
Responsible Party: Principal Investigator, José Herrero Rubí, Principal Investigator and Clinical Professor through the "María Castellano" scolarship (https://orcid.org/0009-0002-9183-6980), IBS Granada
Other Study IDs: CUALIPRIM
Record Dates: First submitted 2025-11-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Age 65 and Older; Polypharmacy; Cronic Lung Disease; Mental Disorder
Keywords: Longitudinality.; Qualitative Research; Health Workforce; Professional-Patient Relations; General Practice
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective To explore and describe the opinions of Primary Health Care chronically ill users regarding being cared for over time by the same reference professional.

To analyze the consequences of workforce instability and the lack of continuity in medical staffing in Primary Health Care centers in Granada.

Design Descriptive observational cross-sectional study using a qualitative methodology. In-depth semi-structured interviews were conducted with users of Primary Health Care centers in Granada.

Setting Primary Health Care in Granada and surrounding rural areas.

Participants Primary Health Care users who attend their Health Centers or Clinics several times a year and have recently experienced a period without a regular family doctor.

Data Collection Tool In-depth interview.

Analysis Qualitative analysis from a phenomenological-ethnographic paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to a physician's patient list that has lacked a regular family doctor for at least 3 of the past 6 months.
* The same list must have been cared for by a single family physician for at least 2 consecutive years in the last 10 years.
* Age 75 or older.
* Presence of a chronic condition requiring medical care at least twice a year (e.g., diabetes, chronic non-cancer pain, heart failure, COPD, mental disorders).
* Use of six or more medications.
* Socioeconomic and social vulnerability.
* Dependence and presence of informal caregivers.

Exclusion criteria:

• Being under 18 years old.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family Care Units (Unidades de Atención Familiar, UAFs) in which the same family physician was assigned for at least six consecutive months and who have subsequently lacked a regular physician for the past six months. Patients with any criteria of chronicity
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Transversal qualitative exploration | Each patient will be interviewed once, after the loss of their long-term assigned primary care physician. Only baseline information will be collected over a period of less than one year, throughout 2024, until study completion.
  Individual semi-structured interviews will be conducted. This format allows for flexibility to accommodate participants' needs and preferences regarding the time and location of the interview (for example, in the participant's own home).
  The interview will begin with an open-ended starter question:
  "What does it mean to you to always be cared for by the same family doctor?"
  Based on the potential themes that may emerge from participants' narratives, a set of research questions has been developed and translated into interview prompts to guide the interviewer. These include:
  Have you noticed any difference in how your health problems are managed when you already know the doctor attending you? Do you think the relationship established with your doctor affects the quality of care you receive? Do you experience any barriers in healthcare when you don't have a regular family doctor? Have you ever withheld a health concern because you didn't know the professional attending you?

CONTACTS AND LOCATIONS:
Overall Officials: José Herrero Rubí, Medicine, Principal Investigator — Servicio Andaluz de Salud - IBS
Locations (2):
- Spain (2):
  - Zaidin Sur Health Centre, Granada, Granada
  - Servicio Andaluz de Salud - IBS, Granada

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the Principal Investigator, JHR. The data are not publicly available as they contain information that could compromise the anonymity of research participants.

DOCUMENTS (2):
  • Study Protocol (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT07320053/Prot_000.pdf
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT07320053/ICF_001.pdf